CLINICAL TRIAL: NCT01016002
Title: A Phase II, Open-label, Single-arm Study of Photodynamic Laser Therapy Using Foscan for Non-curatively-resectable Bile Duct Carcinoma
Brief Title: Single-arm Study of Photodynamic Laser Therapy Using Foscan for Non-curatively-resectable Bile Duct Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Salzburg (Other)
Collaborators: Biolitec Pharma Ltd. (Industry)
Responsible Party: Prof. Frieder Berr, M.D., Department of Internal Medicine I, Paracelsus Medical University Salzburg, Muellner Hauptstrasse 48, 5020, Salzburg, Austria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Foscan 1/2005; EUDRA CT 2005-004866-17
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Non-curative Resectable Bile Duct Carcinoma
MeSH Terms: interventions — temoporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Drug: Temoporfin

INTERVENTIONS:
Drug: Temoporfin — Drug treatment: Temoporfin 0.15 mg/kg body weight, intravenous injection within at least 6 min.
  Laser Treatment: 652nm wavelength; 30 Joules/cm diffusor length ( 200 sec at 150mW/cm diffusor length), within 96 h after Foscan
  Other Names: Foscan; Meso-tetrahydroxyphenyl Chlorin

SUMMARY:
The purpose of this study is to assess efficacy and safety of Foscan (temoporfin) photodynamic therapy in the treatment of locally advanced perihilar bile duct carcinoma without distant metastases.

ELIGIBILITY:
Inclusion Criteria:

* bile duct carcinoma proven by histology in advanced or non-operable stage or tumor extension:

  1. Bismuth type III or IV ( not resectable with R0-margins )
  2. Bismuth type I or II, if resective surgery is contraindicated for old age or poor surgical risk of patient
* sufficient general condition to undergo PDT (Karnofsky status > 30%)
* age > 19 years
* access to common bile duct (either via endoscopy after sphincterotomy or percutaneously after transhepatic drainage),
* informed written consent

Exclusion Criteria:

* porphyria or other diseases exacerbated by light
* known intolerance or allergies to porphyrin derivatives
* a planned surgical procedure within the next 30 days
* coexisting ophthalmic disease likely to require slit lamp examination within the next 30 days
* impaired kidney or liver function (creatinine > 2.5x elevated, INR > 2.2 on vitamin K),
* leukopenia ( WBC < 2000/cmm ) or thrombopenia ( < 50000/cmm ),
* cytotoxic chemotherapy within the past 4 weeks.
* pregnancy ( and safe contraception for 6 months after PDT )
* accompanying/complicating disease with very poor prognosis (expected survival < 6 weeks),
* proven advanced peritoneal carcinomatosis ( PET scan imaging, ascites positive for tumor cells)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Rate of local response and depth of tumoricidal tissue penetration of Foscan-PDT | post treatment

SECONDARY OUTCOMES:
Progression-free survival time, overall survival time | Before first intervention and at months 1, 3, 6, 9, 12, 18 and 24 after intervention
Toxicity using WHO criteria and criteria for local toxicity in the biliary system | Before first intervention and at months 1, 3, 6, 9, 12, 18 and 24 after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Frieder Berr, Prof., MD, Principal Investigator — Department of Internal Medicine I, Paracelsus Medical University Salzburg, Muellner Hauptstrasse 48, 5020, Salzburg, Austria; Lohse A, Prof., MD, Principal Investigator — University Medical Center Hamburg-Eppendorf, Martinistr. 52, 20246 Hamburg, Germany
Locations (2):
- Department of Internal Medicine I, Paracelsus Medical University Salzburg, Salzburg, Salzburg, Austria
- Internal Medicine Dept., University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg, Germany